CLINICAL TRIAL: NCT02015026
Title: Natural History and Tissue Acquisition Study of Adrenocortical Carcinoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140029; 14-C-0029
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-03-02

CONDITIONS: Adrenocortical Carcinoma
Keywords: Biospecimen Repository; Disease Progression Pattern; Specimen Analysis; Genetic Analysis
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

* Adrenocortical carcinoma (ACC) is a rare tumor with an incidence of 1.5 to 2 per million people per year. It has a very poor prognosis with an overall 5-year mortality rate of 75 - 90% and an average survival from the time of diagnosis of 14.5 months.
* The treatment of choice for a localized primary or recurrent tumor is surgical resection.

Patients with recurrent or metastatic disease are infrequently curable by surgery alone.

* As with most solid tumors, chemotherapy options have limited benefit, although platinumbased therapies have response rates of 25 to 30%. To date no targeted therapy has been shown to be of any value in this disease.
* The natural history of ACC can vary greatly with some patients surviving only months while others can live with disease for years. The basis for these differing clinical presentations is not known. While one cannot exclude an immune or other host component as responsible for the diverse clinical courses, it is also possible that there may be a genetic basis for this phenomenon. A bio-specimen repository will be a major step towards more comprehensive studies of this very rare and unusual tumor, and allow us to begin to characterize subgroups within the disease.
* Patients with rare tumors seek expert advice in the management of their care. Dr. Fojo has such expertise and is frequently asked to consult in the care of ACC patients throughout the world. A natural history study would establish a more formal mechanism for such referrals, while allowing the systematic collection of epidemiologic data as well as much needed tumor samples.

Objective:

-To characterize the natural history of adrenocortical cancer, and in the process, collect blood, and tissue samples to study genetic/biochemical pathways involved in the development and progression of adrenocortical cancer (ACC).

Eligibility:

* Patients greater than or equal to 12 years of age with biopsy-proven ACC
* Patients greater than or equal to 12 years of age suspected of having ACC

Design/Schema:

* Patients will be offered clinical consultation with treatment recommendations, including standard of care and clinical trial options. Computed tomography scans of the thorax, abdomen and pelvis will be performed for staging purposes as indicated; occasionally, magnetic resonance imaging will be performed for the visualization of lesions in the liver, spine, or other anatomic sites.
* Medical histories will be documented and patients followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses and hormone production in patients with hormone production as a manifestation of their disease. Tumor growth rates will also be calculated throughout the course of the disease.
* Blood and tumor samples will be obtained at baseline and at follow-up intervals when surgery is indicated. Tumor samples may include samples harvested at other facilities during or prior to enrollment on this trial.
* Genetic and epigenetic analysis of tumors and in selected cases expression array analysis will be performed.

DETAILED DESCRIPTION:
Background:

* Adrenocortical carcinoma (ACC) is a rare tumor with an incidence of 1.5 to 2 per million people per year. It has a very poor prognosis with an overall 5-year mortality rate of 75 - 90% and an average survival from the time of diagnosis of 14.5 months.
* The treatment of choice for a localized primary or recurrent tumor is surgical resection.

Patients with recurrent or metastatic disease are infrequently curable by surgery alone.

* As with most solid tumors, chemotherapy options have limited benefit, although platinumbased therapies have response rates of 25 to 30%. To date no targeted therapy has been shown to be of any value in this disease.
* The natural history of ACC can vary greatly with some patients surviving only months while others can live with disease for years. The basis for these differing clinical presentations is not known. While one cannot exclude an immune or other host component as responsible for the diverse clinical courses, it is also possible that there may be a genetic basis for this phenomenon. A bio-specimen repository will be a major step towards more comprehensive studies of this very rare and unusual tumor, and allow us to begin to characterize subgroups within the disease.
* Patients with rare tumors seek expert advice in the management of their care. A natural history study would establish a more formal mechanism for such referrals, while allowing the systematic collection of epidemiologic data as well as much needed tumor samples.

Objective:

-To characterize the natural history of adrenocortical cancer, and in the process, collect blood, and tissue samples to study genetic/biochemical pathways involved in the development and progression of adrenocortical cancer (ACC).

Eligibility:

* Patients greater than or equal to 12 years of age with biopsy-proven ACC
* Patients greater than or equal to 12 years of age suspected of having ACC

Design/Schema:

* Patients will be offered clinical consultation with treatment recommendations, including standard of care and clinical trial options. Computed tomography scans of the thorax, abdomen and pelvis will be performed for staging purposes as indicated; occasionally, magnetic resonance imaging will be performed for the visualization of lesions in the liver, spine, or other anatomic sites.
* Medical histories will be documented and patients followed throughout the course of their illnesses, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses and hormone production in patients with hormone production as a manifestation of their disease. Tumor growth rates will also be calculated throughout the course of the disease.
* Blood and tumor samples will be obtained at baseline and at follow-up intervals when surgery is indicated. Tumor samples may include samples harvested at other facilities during or prior to enrollment on this trial.
* Genetic and epigenetic analysis of tumors and in selected cases expression array analysis will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients greater than or equal to 12 years of age with biopsy-proven ACC that has been confirmed by the Laboratory of Pathology, NCI.
* Patients greater than or equal to 12 years of age suspected of having ACC. Patients with suspected ACC will undergo baseline workup at the clinical center and be referred for definitive surgical diagnosis and treatment.
* Ability of subject or Legally Authorized Representative to understand and the willingness to sign a written informed consent document.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-12-13; Primary Completion 2015-10-16 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Characterize the natural history of adrenocortical cancer (ACC). Data will include clinical presentation, patterns of disease progression, response or lack of response to therapeutic interventions, disease recurrence and overall survival. | 10 years

SECONDARY OUTCOMES:
Establish a bio-specimen repository for genetic and epigenetic analysis of tumors and in selected cases for expression array analysis by collecting blood, and tissue samples to study the biology of ACC development and progression. | 10 years
Estimate the growth and regression rate constants of tumor treated with standard of care or experimental therapies and correlate with genetic, epigenetic and gene expression profiles | 10 years
Correlate clinical evolution with genetic alterations, DNA methylation patterns and gene expression profiles identified within tumors. | 10 years
Correlate patterns of disease recurrence and impact on progression-free survival and overall survival following a laparoscopic resection or open laparotomy for ACC | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy L Davis, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Terzolo M, Berruti A. Adjunctive treatment of adrenocortical carcinoma. Curr Opin Endocrinol Diabetes Obes. 2008 Jun;15(3):221-6. doi: 10.1097/MED.0b013e3282fdf4c0. PMID 18438168
- [Background] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Background] Stein WD, Yang J, Bates SE, Fojo T. Bevacizumab reduces the growth rate constants of renal carcinomas: a novel algorithm suggests early discontinuation of bevacizumab resulted in a lack of survival advantage. Oncologist. 2008 Oct;13(10):1055-62. doi: 10.1634/theoncologist.2008-0016. Epub 2008 Sep 30. PMID 18827177